CLINICAL TRIAL: NCT03625232
Title: Multi-Center Post-Marketing Study Protocol: (MC-PMS) A Single-arm Open Label Observational Study to Further Document the Safety and Effectiveness of the Epidural Space Verification With the CompuFlo® Epidural Computer Controlled System
Brief Title: Epidural Space Verification With the CompuFlo®
Acronym: MC-PMS
Status: Completed | Type: Observational
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Principal Investigator, Capogna Giorgio, Director EESOA, European e-Learning School in Obstetric Anesthesia
Other Study IDs: EESOA
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Epidural; Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: CompuFlo® Epidural Computer Controlled System — The CompuFlo® Epidural Instrument allows the objective identification of the epidural space by pressure measurement at the needle tip and consequently enables the HCP to perform epidural anesthesia and epidural injections using standard methods. Currently, HCPs rely on their subjective perception to feel a "loss of resistance" when inserting an epidural needle to identify the epidural space. The CompuFlo® Epidural Computer Controlled Anesthesia System has received a CE mark in the European Union and it received 510(k) clearance from the FDA in June 2017.

SUMMARY:
The purpose of this single arm open-label study is to capture additional data that can add to the original COMPASS (CompuFlo® Assessment Study) clinical trial database that supported the 510(k) application, which was given clearance by the FDA on June 9, 2017.

DETAILED DESCRIPTION:
Patients will receive lumbar epidural anesthesia by a HCP, as detailed below. The CompuFlo Epidural System will be utilized only for steps d-g, all other steps are performed in the same way as with the Loss of Resistance Syringe. Refer to User Manual for detailed instructions on how to set up the system.

1. American Society of Anesthesiologists standard monitors will be attached and patients will be placed in a sitting position. Sedation will not be permitted due to potential confounding of the data and/or making it impossible to assess neurological injury/paresthesias during the procedure. Limited Vital signs (blood pressure, apical heart rate, oral temperature, respiration rate) will be obtained and documented in the CRF.
2. Set up the CompuFlo System disposable kit and attach kit to instrument.

   1. Connect the pressure sensor to the ID adapter.
   2. Connect the ID adapter to the CompuFlo instrument.
   3. Connect the external pressure sensor to the filled 20 mL syringe.
   4. Connect the extension tubing to the other end of the pressure sensor.
3. The lumbar area will be disinfected and draped in the usual fashion. The skin in the lumbar area will be locally infiltrated with a local anesthetic solution, according to local practice.
4. The epidural needle will be introduced in the lumbar area to a depth of approximately 3 cm. Insertion to a depth of 3 cm is typical in clinical practice, to avoid accidental epidural space puncture by inserting the needle too deep, while at the same time inserting the needle to a depth at which it will be supported by the tissue.
5. Purge (i.e., prime) the extension tubing connected to the CompuFlo instrument.
6. The CompuFlo extension tubing set will be held at the same vertical height as the puncture level of the epidural needle to calibrate the pressure by depressing the "Zero" button of the CompuFlo® instrument. This will zero the pressure prior to connection of the epidural needle to the extension tubing. The stylet of the epidural needle will be removed and extension tubing will be connected after making the zeroed pressure calibration at the puncture's level.
7. The CompuFlo Epidural Instrument will be set to deliver normal saline at a rate of 0.050 mL/sec during these measurements with an exit-pressure limit not to exceed 120 mm/Hg.
8. The epidural Tuohy needle (18-gauge 3-1/2 inch or any other size) will then be advanced until the pressure readings on the CompuFlo Epidural System indicate position in the epidural space as defined below.

   The following criteria is used to differentiate a True-Loss of Resistance (True-LOR) versus the identification of a False-Loss of Resistance (False-LOR) using the CompuFlo Epidural Instrument:

   A True-LOR defined as:

   An increase in pressure followed by a sudden and sustained (> 5 seconds) drop in pressure (typically greater than 50% of the maximum pressure), resulting in the formation of a "low and stable pressure plateau"

   A False-LOR defined as:

   An increase of pressure followed by a drop in pressure (typically less than 50% of the maximum pressure) that is either not sustained or inconclusive of representing a "low and stable pressure plateau"

   -If the pressure rapidly increases after a drop of pressure this is identified as a False-Loss of Resistance and the operator may elect to continue to advance the needle.

   A Inconclusive-LOR defined as:

   -If the pressure does not increase or is deemed to be inconclusive (Undeterminable) loss of resistance the operator should withdraw the needle and/or redirect the needle. This will be considered an Inconclusive-LOR (I-LOR)

   Number of attempts* will be defined and measured as follows:
   1. Number of needle withdrawals and reinsertions at the same interspace
   2. Number of needle withdrawals and reinsertions at a different interspace
   3. Number needle redirections in case of bone contact
   4. Number needle redirections due to operator's uncertainty of needle location (inconclusive or undeterminable) loss of resistance *Definitions: 1 and 2: the needle is completely withdrawn and reinserted from the skin 3 an 4: the needle is redirected and/or partially withdrawn to allow redirection within the tissues of the chosen interspace

   NOTE: When every a drop of pressure occurs during the advancement** of a needle it is critical that the operator simultaneously STOP ALL NEEDLE MOVEMENT to determine if any further pressure changes will occur based on the position of the needle.

   ** NOTE: The CompuFlo-Epidural Instrument is a highly accurate device capable of recording all information continuously and precisely. Be aware that the operator can introduce pressure artifacts to the data recordings if imprecise needle movements are used, such as a rapid advancement and/or rapid withdrawals of the needle not representative of standard clinical needle movements. The pressure wave-form slope of the curve is impacted by imprecise needle movements. Therefore, slow deliberate needle movements are recommended.

   The readings on the CompuFlo Epidural Instrument that correlate with correct epidural space identification (True-LOR) based on the previous trial conducted by Ghelber et al. consist of the following criteria:

   After documenting the significant drop in pressure for at least 5 seconds, with no further needle movement:
   1. Record an additional 5 seconds of pressure data, with the motor running to identify the formation of a low and stable low pressure plateau, (typically greater than 50% of the maximum pressure).
   2. Press STOP and continue to record pressure for 5 additional seconds, after the motor has stopped, while the needle is still in the epidural space to record the EPIDURAL SPACE PRESSURE.
   3. To investigate possible waveform patterns which may confirm the entrance of the needle in the epidural space, after these additional 5 seconds, request that patient either "cough" and record the epidural pressure (PRESSURE AFTER COUGH) or perform a 2-3 seconds Valsalva maneuver and record the epidural pressure at the apex of the maneuvre (PRESSURE AFTER VALSALVA) .
   4. Once the CompuFlo® procedure is complete, Press END PROCEDURE to ensure that the data file is properly saved. Then Press YES to terminate procedure. NOTE: Avoiding this step will lead to the loss and/or corruption of data file.

   These steps provide a secondary means of verification of the epidural space. If the correct position of the epidural Tuohy needle in the epidural space (as indicated by the readings on the CompuFlo® Epidural System) can NOT be obtained or dye injection indicates incorrect position or an epidural catheter cannot be advanced into the epidural space, then the epidural Tuohy needle will be withdrawn or redirected and a new attempt of epidural Tuohy needle insertion and identification of the epidural space with the CompuFlo® Epidural System will begin. Alternatively, the HCP and/or anesthesiologist can choose to completely remove the epidural Tuohy needle and insert at a new puncture site and a new attempt of epidural Tuohy needle insertion and identification of the epidural space with the CompuFlo® Epidural System will begin. The local investigator may decide after a number of failed recorded attempts to suspend the procedure. Then, epidural anesthesia with the CompuFlo® Epidural System will be considered unsuccessful and the patient will be converted to other forms of analgesia.
9. After successful epidural space identification, the CompuFlo® Epidural System will be disconnected from the epidural needle and an epidural catheter will be advanced 3-5cm into the epidural space, or injection will proceed according to standard medical practice if there is no introduction of an epidural catheter.

   4. After removal of the epidural needle and securing of the epidural catheter, an epidural test dose consisting - in the case of epidural labor analgesia - of the therapeutic dose, if a low concentration local anesthetic solution is used (e.g., bupivacaine 0.0625%) or a 3 mL epidural test dose (lidocaine 15 mg/mL with epinephrine 5 mcg/mL), if a high concentration (e.g., bupivacaine 0.25, 0.125%) is used, will be manually infused to rule out intrathecal or intravascular catheter position for those procedures where test dose is considered standard medical practice.
10. Epidural anesthesia or any medical treatment according to HCP order will then be delivered by dosing the epidural catheter with a local anesthetic/medication of the HCP's choice and a volume of their choice that should conform to that described in the local anesthetic's labeling.

For a woman in labor, successful performance of epidural procedure will be defined as the occurrence of analgesia assessed by Visual Analogue Pain Scale (VAPS), after a predetermined period of time from the epidural loading dose. (Ex., a VAPS < 10 at 20 min.) For other epidural procedures, successful performance of an epidural procedure will be defined as a loss of sensation to cold in at least in one dermatome. Alternatively, for subjects not in a labor while undergoing epidural procedures that are assisted by fluoroscopy, successful performance will be defined as correct spread of dye in the epidural space, as judged by an independent HCP.

At that time limited vital signs (blood pressure, apical heart rate, oral temperature, respiration rate) will be obtained and documented in the CRF.

In case of a unilateral block, the HCP will be permitted to manipulate the catheter at their discretion (e.g., withdraw the catheter) and re-dose the catheter. In such case, another assessment of loss of sensation to cold as described above will be permitted 30 min after catheter re-dosing to assess whether epidural anesthesia was successful (same criteria as above).

If analgesia for women in labor or one dermatome for other patients cannot be established, epidural procedure/anesthesia will be considered unsuccessful and the patient will receive analgesia or anesthesia at the discretion of the HCP.

The number of attempts (needle redirection and reinsertions) will be recorded.

For those sites performing fluoroscopy/dye injection, an indication of incorrect spread of the dye will be considered failure.

Within thirty minutes after dosing the epidural catheter, a blinded investigator will assess the patient for sensory and motor blockade.

Concomitant medication, including conversion to general anesthesia, along with any adverse events will also be recorded.

All of these assessments will be recorded in the source documents and on the appropriate CRFs.

After the completion of the epidural procedure, the physician will complete the Compuflo Assessment Score Questionnaire (Section 9.4) to assess the agreement between the physician' s reported sensation and the variation of pressure given by the CompuFlo® during the needle tracking from its insertion until the identification of the epidural space.

Any occurrence of accidental dural puncture with the Tuohy needle during the epidural procedure assisted by Compuflo will be recorded on the data sheet.

The occurrence of Post Dural Puncture Headache (PDPH) will be also recorded. PDPH will be defined according to the Classification Committee of The International Headache Society (https://www.ichd-3.org/7-headache-attributed-to-non-vascular-intracranial-disorder/7-2-headache-attributed-to-low-cerebrospinal-fluid-pressure/7-2-1-post-dural-puncture-headache/)

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age at screening, but has not had his/her 91st birthday.
* The subject is required to have epidural procedure implemented as part of their standard medical treatment according to Principal Investigator assessment.
* The subject and/or legally authorized person/representative is willing to undergo the Informed Consent process prior to enrollment into this study.
* The subject is willing to participate in this study for at least 30 days after the epidural procedure implementation.
* The subject is willing to participate in this study for at least 3 days after the procedure.

Exclusion Criteria:

* Contraindications for epidural procedure / anesthesia (circumstances where the risks associated with epidural procedures are higher than usual. These circumstances are, but not limited to, anatomical abnormalities, such as spina bifida or scoliosis, infection at or near the site of insertion, allergy to the anesthetic or intended drug, uncorrected hypovolemia, increased intracranial pressure etc.).
* Patients presenting for emergency C-section or other emergencies.
* Exclusive use of other treatments such as intravenous analgesia with opioids.
* Prior back surgery in lumbar area that would prevent epidural access.
* Preexisting neurological deficit that would interfere with dermatome identification.
* The subject observed seizure within 7 days prior to study enrollment.
* Presumed and/or confirmed septic embolus.
* The subject has a skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) in their lumbar region greater than 4 cm2.
* The subject previously participated in another investigational drug or device trial within the preceding 4 weeks.
* Severe co-existing or terminal systemic disease that limits life expectancy or may interfere with study procedures.
* The subject is otherwise determined by the Investigator to be medically unsuitable for participation in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for this study will consist of up to 800 adult subjects between the ages of 18 and 90 (had 18th birthday and had not had their 91st birthday - except for State of Alabama where legal consent for adults is age of 19), of any ethnic background, for whom an epidural procedure is indicated according to their HCP. The subject will meet all the inclusion criteria, have none of the exclusion criteria, give their written Informed Consent to participate in this clinical study after undergoing informed consent process, In the event that a subject's ability to comprehend and communicate is compromised (per the discretion of the Principal Investigator), a legal representative may discuss the study, agree on participation and sign the ICF, on behalf of the subject.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Visual Analogue Pain Scale | 20 minutes
  Number of patients with Visual Analogue Pain Scale (VAPS ) score (0 = non pain; 100 = maximum pain) less than 20 after 20/30 minutes from the epidural analgesic loading dose or for those patients for whom fluoroscopy is performed: Number of patients having correct spread of dye in the epidural space as observed by fluoroscopy
Epidural identification | 15 minutes
  To Identify and differentiate True-LOR vs. False-LOR and/or Inconclusive-LOR during ES identification by using the Compuflo Epidural Instrument recordings of pressure (delta, mmHg)
  A True-LOR defined as:
  An increase in pressure followed by a sudden and sustained (> 5 seconds) drop in pressure (mmHg) resulting in the formation of a low and stable pressure plateau
  A False-LOR defined as:
  An increase of pressure (mmHg) followed by a drop in pressure that is either not sustained or inconclusive of representing a "low and stable pressure plateau" If the pressure (mmHg) rapidly increases after a drop of pressure this is identified as a False-Loss of Resistance and the operator may elect to continue to advance the needle.
Complications | 36 hours
  Number of patients having inadvertent dural punture Number of patients having post dural punture headache

SECONDARY OUTCOMES:
Physician Concordance Index | 24 hours
  The agreement between the physician's reported sensation and the variation of pressure given by the CompuFlo® during the needle tracking from its insertion until the identification of the epidural space will be evaluated by using a 5 poin Likert scale
  1 2 3 4 5 (From Strongly disagree to Strongly agree) Completed immediately after each procedure by the physician who performed block
Secondary Epidural Veriification | 15 minutes
  After documenting the significant drop in pressure (mmHg) for at least 5 seconds, with no further needle movement:
  1. additional 5 seconds of pressure data (mmHg) will be recorded to identify the formation of a low and stable low pressure plateau
  2. Compuflo motor will be stopped and the pressure will be recorded for 5 additional seconds, while the needle is still in the epidural space to record the EPIDURAL SPACE PRESSURE (mmHg).
  3. The patients will be requested either to cough and the epidural pressure will be recorded (PRESSURE AFTER COUGH, mmHg)) or to perform a 2-3 seconds Valsalva maneuver andthe epidural pressure at the apex of the maneuvre (PRESSURE AFTER VALSALVA, mmHg) will be recorded .

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (11):
- University Hospital Leuven, Leuven, Belgium
- Alemanno Hospital, Santiago, Chile
- Klinik und Poliklinik für Anästhesiologie, Würzburg, Germany
- Italy (6):
  - Casa di Cura Gibiino, Università di Catania, Catania
  - Careggi Hospital, Florence
  - Casa Sollievo Sofferenza, S Giovanni Rotondo, Foggia
  - Clinica Mangiagalli, Milan
  - Ospedale Buccheri La Ferla, Palermo
  - Città di Roma Hospital, Rome
- Madrid University Hospital, Madrid, Spain
- Frimley Park Hospital, Frimley, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Capogna G, Coccoluto A, Capogna E, Del Vecchio A. Objective Evaluation of a New Epidural Simulator by the CompuFlo(R) Epidural Instrument. Anesthesiol Res Pract. 2018 Jun 26;2018:4710263. doi: 10.1155/2018/4710263. eCollection 2018. PMID 30046305